CLINICAL TRIAL: NCT02896153
Title: Current Situation on the Consumption of Hypnotic Substances at the Pharmacy
Acronym: HYPNOSIS
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC14_0421
Record Dates: First submitted 2016-08-05; First posted 2016-09-12 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Substances Used for a Hypnotic Purpose
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Adult population going to a pharmacy: Adult population going to a pharmacy will be asked to complete a questionnaire.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire

SUMMARY:
In France, consumption of hypnotic drugs is high. In this context, and given the planned regulatory modifications, it seems essential to make an inventory of the consumption of drugs taken for a hypnotic purpose. This study aims to identify the substances (medical or not) used for a hypnotic purpose in the adult population going to a pharmacy.

ELIGIBILITY:
Inclusion Criteria:

* Adult going to the pharmacy and who accepts to complete the questionnaire

Exclusion Criteria:

* Minor
* Who is not able to complete a questionnaire
* Who does not accept to complete the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult going to a pharmacy
Sampling Method: Non-Probability Sample
Enrollment: 657 (Actual)
Dates: Start 2014-12; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The name of the substance (medical or not) used for a hypnotic purpose | One day